CLINICAL TRIAL: NCT04615780
Title: Effectiveness of Green Tea Mouthwash on the Oral Health Status in Oral Cancer Patients: A Single-blind Randomized Clinical Trial and a CONSORT-compliant Article
Brief Title: Green Tea Mouthwash on the Oral Health Status in Oral Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10717
Record Dates: First submitted 2020-10-27; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms | interventions — Mouthwashes; Tea

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to 2 groups: mouthwash with green tea (intervention) group or tap water (control) group. The intervention group rinsed the mouth with 100 ml green tea solution for 60 seconds at least twice daily, and the control group rinsed the mouth with 100 ml tap water for 60 seconds at least twice daily.
Masking Description: Because of the nature of the intervention, only the data analyst was blinded to the meaning of the group assignment code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mouthwash with green tea group (Experimental): The intervention group rinsed the mouth with 100 ml green tea solution for 60 seconds at least twice daily.
  Interventions: Other: mouthwash with green tea
- mouthwash with tap water group (Placebo Comparator): The control group rinsed the mouth with 100 ml tap water for 60 seconds at least twice daily.
  Interventions: Other: mouthwash with tap water group

INTERVENTIONS:
Other: mouthwash with green tea — All patients received instructions for using the Bass brushing method to brush their teeth with a soft small-headed toothbrush. The intervention group rinsed the mouth with 100 ml green tea solution for 60 seconds at least twice daily. For the preparation of the green tea mouthwash, green tea solution was made with 5 g (1 teaspoon) of green tea powder dissolved in 100 ml water to produce 5% green tea mouthwash, as described in a previous study (Eshghpour, et al., 2013). The green tea powder was ground from Camelia sinensis leaves and regularly provided by the researcher. The green tea solution is made for a single use and remade before rinsing each time. When patients return to the outpatient monthly, the researcher first confirms patients' compliance, then assists with solving difficulties and gives encouragement.
  Arms: mouthwash with green tea group
Other: mouthwash with tap water group — All patients received instructions for using the Bass brushing method to brush their teeth with a soft small-headed toothbrush. The control group rinsed the mouth with 100 ml tap water for 60 seconds at least twice daily.
  Arms: mouthwash with tap water group

SUMMARY:
Objectives: To evaluate the effectiveness of green tea mouthwash on the oral health status (OHS) in oral cancer patients undergoing anticancer treatment.

Materials and methods: This was a prospective, single-blind, randomized, controlled trial. Patients were randomly assigned to 2 groups: mouthwash with green tea (intervention) group or tap water (control) group. The intervention group rinsed the mouth with 100 ml green tea solution for 60 seconds at least twice daily, and the control group rinsed the mouth with 100 ml tap water for 60 seconds at least twice daily. The primary outcome was OHS, which was evaluated according to the Oral Assessment Guide and measured at seven time points by the same researcher. Time 0 (T0) corresponded to baseline, and Time 1-6 (T1-T6) corresponded to monthly outpatient follow-ups until six months.

ELIGIBILITY:
Inclusion Criteria:

* patients who were > 20 years
* newly diagnosed with oral cancer by a physician
* just received oral surgery and follow-up with or without chemotherapy or radiation therapy.

Exclusion Criteria:

* patients with mental illness
* an acute and a severe illness status
* no teeth in the whole mouth
* the ability of mouth opening less than 1 cm.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
oral health status (OHS) | Time 0 (T0) corresponded to baseline
  Patients' oral health status (OHS) was assessed according to the Oral Assessment Guide (OAG) by the same researcher. The OAG consists of eight items: voice, swallow, lips, tongue, saliva, mucous membranes, gingiva and teeth or dentures. Each item is rated by a grading of 1 (normal) to 3 (severe). Sum scores between 8-24 points and a higher score indicate poorer OHS.
oral health status (OHS) | Time 1(T1) corresponded to the 1 month after recruitment.
  Patients' oral health status (OHS) was assessed according to the Oral Assessment Guide (OAG) by the same researcher. The OAG consists of eight items: voice, swallow, lips, tongue, saliva, mucous membranes, gingiva and teeth or dentures. Each item is rated by a grading of 1 (normal) to 3 (severe). Sum scores between 8-24 points and a higher score indicate poorer OHS.
oral health status (OHS) | Time 2(T2) corresponded to the 2nd month after recruitment.
  Patients' oral health status (OHS) was assessed according to the Oral Assessment Guide (OAG) by the same researcher. The OAG consists of eight items: voice, swallow, lips, tongue, saliva, mucous membranes, gingiva and teeth or dentures. Each item is rated by a grading of 1 (normal) to 3 (severe). Sum scores between 8-24 points and a higher score indicate poorer OHS.
oral health status (OHS) | Time 3(T3) corresponded to the 3th month after recruitment.
  Patients' oral health status (OHS) was assessed according to the Oral Assessment Guide (OAG) by the same researcher. The OAG consists of eight items: voice, swallow, lips, tongue, saliva, mucous membranes, gingiva and teeth or dentures. Each item is rated by a grading of 1 (normal) to 3 (severe). Sum scores between 8-24 points and a higher score indicate poorer OHS.
oral health status (OHS) | Time 4(T4) corresponded to the 4th month after recruitment.
  Patients' oral health status (OHS) was assessed according to the Oral Assessment Guide (OAG) by the same researcher. The OAG consists of eight items: voice, swallow, lips, tongue, saliva, mucous membranes, gingiva and teeth or dentures. Each item is rated by a grading of 1 (normal) to 3 (severe). Sum scores between 8-24 points and a higher score indicate poorer OHS.
oral health status (OHS) | Time 5(T5) corresponded to the 5th month after recruitment.
  Patients' oral health status (OHS) was assessed according to the Oral Assessment Guide (OAG) by the same researcher. The OAG consists of eight items: voice, swallow, lips, tongue, saliva, mucous membranes, gingiva and teeth or dentures. Each item is rated by a grading of 1 (normal) to 3 (severe). Sum scores between 8-24 points and a higher score indicate poorer OHS.
oral health status (OHS) | Time 6(T6) corresponded to the 6th month after recruitment.
  Patients' oral health status (OHS) was assessed according to the Oral Assessment Guide (OAG) by the same researcher. The OAG consists of eight items: voice, swallow, lips, tongue, saliva, mucous membranes, gingiva and teeth or dentures. Each item is rated by a grading of 1 (normal) to 3 (severe). Sum scores between 8-24 points and a higher score indicate poorer OHS.

CONTACTS AND LOCATIONS:
Locations (1):
- Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liao YC, Hsu LF, Hsieh LY, Luo YY. Effectiveness of green tea mouthwash for improving oral health status in oral cancer patients: A single-blind randomized controlled trial. Int J Nurs Stud. 2021 Sep;121:103985. doi: 10.1016/j.ijnurstu.2021.103985. Epub 2021 May 25. PMID 34186380